CLINICAL TRIAL: NCT06602544
Title: Preventing Freezing of Gait in Parkinson's Disease Using Soft Robotic Apparel
Brief Title: Robotic Apparel to Prevent Freezing of Gait in Parkinson Disease
Acronym: XF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Michael J Fox Foundation for Parkinson Research (Unknown); Boston University (Other)
Responsible Party: Principal Investigator, Conor Walsh, Professor, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#24-0986; 024589 (Other Grant/Funding Number: Michael J Fox Foundation)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson Disease; Freezing-of-gait; Wearable Robot; Soft Robotics; Gait; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-visit ambulatory activities with soft robotic apparel (Experimental): Participants will engage in ambulatory activities (i.e. straight-line walking, turning) with and without the assistance of robotic apparel, performed across multiple visits under various freezing-of-gait (FoG) provoking scenarios
  Interventions: Device: Robotic Apparel

INTERVENTIONS:
Device: Robotic Apparel — A robotic apparel system is a portable, lightweight textile-based wearable robot that is worn around the waist and thighs. The apparel provides assistive flexion moment about the hip joint during the swing phase of gait by spooling in a cable that connects the thigh wraps to the front of the waist belt. Inertial measurement units embedded in the thigh wraps are used to control the timing of the robotic apparel assistance. Robotic apparel assistance magnitude is delivered as a small percentage of the bodyweight of the wearer.

SUMMARY:
Freezing-of-gait (FoG) in Parkinson Disease (PD) is one of the most vivid and disturbing gait phenomena in neurology. Often described by patients as a feeling of "feet getting glued to the floor," FoG is formally defined as a "brief, episodic absence or marked reduction of forward progression of the feet despite the intention to walk." This debilitating gait phenomena is very common in PD, occurring in up to 80% of individuals with severe PD. When FoG arrests walking, serious consequences can occur such as loss of balance, falls, injurious events, consequent fear of falling, and increased hospitalization. Wearable robots are capable of augmenting spatiotemporal gait mechanics and are emerging as viable solutions for locomotor assistance in various neurological populations. For the proposed study, our goal is to understand how low force mechanical assistance from soft robotic apparel can best mitigate gait decline preceding a freezing episode and subsequent onset of FoG by improving spatial (e.g. stride length) and temporal features (e.g. stride time variability) of walking. We hypothesize that the ongoing gait-preserving effects can essentially minimize the accumulation of motor errors that lead to FoG. Importantly, the autonomous assistance provided by the wearable robot circumvents the need for cognitive or attentional resources, thereby minimizing risks for overloading the cognitive systems -- a known trigger for FoG, thus enhancing the repeatability and robustness of FoG-preventing effects.

DETAILED DESCRIPTION:
Wearable robots are capable of augmenting spatiotemporal gait mechanics and are emerging as viable solutions for locomotor assistance in various neurological populations. Given the breakdown of spatiotemporal gait parameters prior to onset of FoG, we aim to understand how the use of mechanical assistance from a soft robotic apparel can best mitigate gait decline preceding a freezing episode, and subsequent onset of FoG through a multi-day proof-of-concept study. In Aim 1, we will determine the biomechanical mechanisms underpinning the effects of robotic apparel on FoG. We posit that robotic apparel will prevent FoG by supporting natural gait biomechanics and reducing motor errors and gait degradation (i.e., increase stride length, decrease stride variability) known to precede freezing. In Aim 2, we will quantify the impact of robotic apparel in preventing FoG in PD under a variety of walking conditions in a series of controlled laboratory-based experiments. We hypothesize that robotic apparel will be effective in preventing FoG as evidenced by lower percent time spent freezing and lower FoG severity ratio scores (IMU data, video annotation) during walking and turning, resulting in farther walking distances (2-Minute Walk Test) compared to unassisted walking, repeatable across days of testing. Additionally, we hypothesize that robotic apparel will be effective in preventing FoG across various walking contexts (i.e., walking in open spaces, turning, dual-tasking and medication on/off). In Aim 3, we will examine proof-of-concept of robotic apparel to prevent FoG in the home/community during walking, under FoG provoking conditions. We hypothesize that robotic apparel will be effective in preventing FoG, compared to unassisted walking, as evidenced by lower percent time spent freezing and lower FoG severity ratio scores (IMU data, video annotation) during walking in the home/community, including conditions that trigger FoG (e.g., personalized FoG "hotspots).

The study will utilize a soft robotic apparel that has previously shown to demonstrate robust, gait-preserving benefits and FoG prevention in a single-subject repeated measures case study. To examine the effectiveness of the intervention using our robotic apparel, this 9-visit study will collect data on amount of time spent freezing, spatiotemporal gait measures, clinical measures, and patient perspectives on the device during different standardized assessments and freeze-provoking activities across multiple environments (i.e. home, lab) and medication states (on, relative off) with and without the robotic apparel assistance.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* Self-reported Freezing of Gait due to PD
* Score of 21 or higher on the cognitive screening test (Montreal Cognitive Assessment Score (MoCA))
* Independent ambulation (with or without an assistive device, no physical assistance) for at least 20 meters
* Able to understand, communicate, and be understood by study staff
* Provide HIPAA Authorization to allow communication with the participant's treating physician/provider for medical clearance (if deemed necessary by study clinical team) to verify self-reported medical history (if deemed necessary by study clinical team)
* Provide informed consent
* Ability to participate in 8 research study visits

Exclusion Criteria:

* More than 2 falls in the previous month, as a result of gait impairment (may enroll under clinician discretion)
* Major surgery in the last 6 months that interferes with walking (may enroll under clinician discretion)
* Gait deficits due to missing limbs
* Experience chronic pain that interferes with walking ability (may enroll under clinician discretion)
* Serious co-morbidities (unrelated to gait impairment) that may interfere with ability to participate in research (e.g. cardiovascular, neurological, skin, and vascular conditions such as acute, ongoing/unmanaged deep vein thrombosis)
* No observable freezing-of-gait

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in percent time spent freezing | Visit 4 (within 6 months after enrollment)
  Percent time spent freezing refers to cumulative duration spent freezing divided by the total duration of the task, expressed as percentage. Change in this outcome measure refers to the difference in percent time spent freezing during activities with and without assistance of robotic apparel.
Change in percent time spent freezing | Visit 5 (within 6 months after enrollment)
  Percent time spent freezing refers to cumulative duration spent freezing divided by the total duration of the task, expressed as percentage. Change in this outcome measure refers to the difference in percent time spent freezing during activities with and without assistance of robotic apparel.
Change in percent time spent freezing | Visit 6 (within 6 months after enrollment)
  Percent time spent freezing refers to cumulative duration spent freezing divided by the total duration of the task, expressed as percentage. Change in this outcome measure refers to the difference in percent time spent freezing during activities with and without assistance of robotic apparel.
Change in percent time spent freezing | Visit 7 (within 6 months after enrollment)
  Percent time spent freezing refers to cumulative duration spent freezing divided by the total duration of the task, expressed as percentage. Change in this outcome measure refers to the difference in percent time spent freezing during activities with and without assistance of robotic apparel.
Change in percent time spent freezing | Visit 8 (within 6 months after enrollment)
  Percent time spent freezing refers to cumulative duration spent freezing divided by the total duration of the task, expressed as percentage. Change in this outcome measure refers to the difference in percent time spent freezing during activities with and without assistance of robotic apparel.
Change in percent time spent freezing | Visit 9 (within 6 months after enrollment)
  Percent time spent freezing refers to cumulative duration spent freezing divided by the total duration of the task, expressed as percentage. Change in this outcome measure refers to the difference in percent time spent freezing during activities with and without assistance of robotic apparel.
Change in stride length | Visit 4 (within 6 months after enrollment)
  Stride length is the Euclidian distance between a point at heel strike at the beginning of gait cycle and a point at heel strike at the subsequent gait cycle. Change in this outcome measure refers to difference in stride length during activities with and without assistance of robotic apparel.
Change in stride length | Visit 5 (within 6 months after enrollment)
  Stride length is the Euclidian distance between a point at heel strike at the beginning of gait cycle and a point at heel strike at the subsequent gait cycle. Change in this outcome measure refers to difference in stride length during activities with and without assistance of robotic apparel.
Change in stride length | Visit 6 (within 6 months after enrollment)
  Stride length is the Euclidian distance between a point at heel strike at the beginning of gait cycle and a point at heel strike at the subsequent gait cycle. Change in this outcome measure refers to difference in stride length during activities with and without assistance of robotic apparel.
Change in stride length | Visit 7 (within 6 months after enrollment)
  Stride length is the Euclidian distance between a point at heel strike at the beginning of gait cycle and a point at heel strike at the subsequent gait cycle. Change in this outcome measure refers to difference in stride length during activities with and without assistance of robotic apparel.
Change in stride length | Visit 8 (within 6 months after enrollment)
  Stride length is the Euclidian distance between a point at heel strike at the beginning of gait cycle and a point at heel strike at the subsequent gait cycle. Change in this outcome measure refers to difference in stride length during activities with and without assistance of robotic apparel.
Change in stride length | Visit 9 (within 6 months after enrollment)
  Stride length is the Euclidian distance between a point at heel strike at the beginning of gait cycle and a point at heel strike at the subsequent gait cycle. Change in this outcome measure refers to difference in stride length during activities with and without assistance of robotic apparel.

SECONDARY OUTCOMES:
Change in freezing-of-gait ratio | Visit 4 (within 6 months after enrollment)
  Freezing-of-gait ratio refers to the ratio between total power in the 3-8Hz band and the total power in the 0.5-3Hz band in the shank inertial measurement units. Change in this outcome measure refers to difference in freezing-of-gait ratio during activities with and without assistance of robotic apparel.
Change in freezing-of-gait ratio | Visit 5 (within 6 months after enrollment)
  Freezing-of-gait ratio refers to the ratio between total power in the 3-8Hz band and the total power in the 0.5-3Hz band in the shank inertial measurement units. Change in this outcome measure refers to difference in freezing-of-gait ratio during activities with and without assistance of robotic apparel.
Change in freezing-of-gait ratio | Visit 6 (within 6 months after enrollment)
  Freezing-of-gait ratio refers to the ratio between total power in the 3-8Hz band and the total power in the 0.5-3Hz band in the shank inertial measurement units. Change in this outcome measure refers to difference in freezing-of-gait ratio during activities with and without assistance of robotic apparel.
Change in freezing-of-gait ratio | Visit 7 (within 6 months after enrollment)
  Freezing-of-gait ratio refers to the ratio between total power in the 3-8Hz band and the total power in the 0.5-3Hz band in the shank inertial measurement units. Change in this outcome measure refers to difference in freezing-of-gait ratio during activities with and without assistance of robotic apparel.
Change in freezing-of-gait ratio | Visit 8 (within 6 months after enrollment)
  Freezing-of-gait ratio refers to the ratio between total power in the 3-8Hz band and the total power in the 0.5-3Hz band in the shank inertial measurement units. Change in this outcome measure refers to difference in freezing-of-gait ratio during activities with and without assistance of robotic apparel.
Change in freezing-of-gait ratio | Visit 9 (within 6 months after enrollment)
  Freezing-of-gait ratio refers to the ratio between total power in the 3-8Hz band and the total power in the 0.5-3Hz band in the shank inertial measurement units. Change in this outcome measure refers to difference in freezing-of-gait ratio during activities with and without assistance of robotic apparel.
Change in 2-Minute Walk Test Distance | Visit 5 (within 6 months after enrollment)
  2-Minute Walk Test distance refers to the farthest distance covered during 2 minutes of walking. Change in this outcome measure refers to difference in the 2-Minute Walk Test distance with and without assistance of robotic apparel.
Change in 2-Minute Walk Test Distance | Visit 6 (within 6 months after enrollment)
  2-Minute Walk Test distance refers to the farthest distance covered during 2 minutes of walking. Change in this outcome measure refers to difference in the 2-Minute Walk Test distance with and without assistance of robotic apparel.
Change in 2-Minute Walk Test Distance | Visit 7 (within 6 months after enrollment)
  2-Minute Walk Test distance refers to the farthest distance covered during 2 minutes of walking. Change in this outcome measure refers to difference in the 2-Minute Walk Test distance with and without assistance of robotic apparel.
Change in 2-Minute Walk Test Distance | Visit 8 (within 6 months after enrollment)
  2-Minute Walk Test distance refers to the farthest distance covered during 2 minutes of walking. Change in this outcome measure refers to difference in the 2-Minute Walk Test distance with and without assistance of robotic apparel.
Change in 2-Minute Walk Test Distance | Visit 9 (within 6 months after enrollment)
  2-Minute Walk Test distance refers to the farthest distance covered during 2 minutes of walking. Change in this outcome measure refers to difference in the 2-Minute Walk Test distance with and without assistance of robotic apparel.
Change in range of motion | Visit 4 (within 6 months after enrollment)
  Range of motion refers to the range (difference in maximum and minimum) of sagittal plane motion of the hip, knee, and ankle joints throughout a gait cycle. Change in this outcome measure refers to difference in the hip, ankle, and knee range-of-motion during activities with and without assistance of robotic apparel.
Change in cadence | Visit 4 (within 6 months after enrollment)
  Cadence refers to the number of steps or strides taken per minute. Change in this outcome measure refers to difference in the cadence during activities with and without assistance of robotic apparel.
Change in cadence | Visit 5 (within 6 months after enrollment)
  Cadence refers to the number of steps or strides taken per minute. Change in this outcome measure refers to difference in the cadence during activities with and without assistance of robotic apparel.
Change in cadence | Visit 6 (within 6 months after enrollment)
  Cadence refers to the number of steps or strides taken per minute. Change in this outcome measure refers to difference in the cadence during activities with and without assistance of robotic apparel.
Change in cadence | Visit 7 (within 6 months after enrollment)
  Cadence refers to the number of steps or strides taken per minute. Change in this outcome measure refers to difference in the cadence during activities with and without assistance of robotic apparel.
Change in cadence | Visit 8 (within 6 months after enrollment)
  Cadence refers to the number of steps or strides taken per minute. Change in this outcome measure refers to difference in the cadence during activities with and without assistance of robotic apparel.
Change in cadence | Visit 9 (within 6 months after enrollment)
  Cadence refers to the number of steps or strides taken per minute. Change in this outcome measure refers to difference in the cadence during activities with and without assistance of robotic apparel.
Change in stride time variability | Visit 4 (within 6 months after enrollment)
  Stride time variability refers to the difference in the coefficient of variance of stride time in each activity bout. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.
Change in stride time variability | Visit 5 (within 6 months after enrollment)
  Stride time variability refers to the difference in the coefficient of variance of stride time in each activity bout. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.
Change in stride time variability | Visit 6 (within 6 months after enrollment)
  Stride time variability refers to the difference in the coefficient of variance of stride time in each activity bout. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.
Change in stride time variability | Visit 7 (within 6 months after enrollment)
  Stride time variability refers to the difference in the coefficient of variance of stride time in each activity bout. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.
Change in stride time variability | Visit 8 (within 6 months after enrollment)
  Stride time variability refers to the difference in the coefficient of variance of stride time in each activity bout. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.
Change in stride time variability | Visit 9 (within 6 months after enrollment)
  Stride time variability refers to the difference in the coefficient of variance of stride time in each activity bout. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.
Change in peak foot-to-floor angle | Visit 4 (within 6 months after enrollment)
  Peak foot-to-floor angle refers to the maximum angle of the foot relative to ground as the foot dorsiflexes at heel strike, measured by the foot inertial measurement unit. Change in this outcome measure refers to difference in the stride time variability during activities with and without assistance of robotic apparel.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ellis, PT, PhD, Principal Investigator — Boston University; Conor J Walsh, PhD, Principal Investigator — Harvard University
Locations (2):
- United States (2):
  - Harvard Science and Engineering Complex, Allston, Massachusetts
  - Boston University Sargent College of Health and Rehabilitation Sciences, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ziegler K, Schroeteler F, Ceballos-Baumann AO, Fietzek UM. A new rating instrument to assess festination and freezing gait in Parkinsonian patients. Mov Disord. 2010 Jun 15;25(8):1012-8. doi: 10.1002/mds.22993. PMID 20310009
- [Background] Ehgoetz Martens KA, Shine JM, Walton CC, Georgiades MJ, Gilat M, Hall JM, Muller AJ, Szeto JYY, Lewis SJG. Evidence for subtypes of freezing of gait in Parkinson's disease. Mov Disord. 2018 Jul;33(7):1174-1178. doi: 10.1002/mds.27417. PMID 30153383
- [Background] Plotnik M, Giladi N, Hausdorff JM. Is freezing of gait in Parkinson's disease a result of multiple gait impairments? Implications for treatment. Parkinsons Dis. 2012;2012:459321. doi: 10.1155/2012/459321. Epub 2012 Jan 12. PMID 22288021
- [Background] Nieuwboer A, Giladi N. Characterizing freezing of gait in Parkinson's disease: models of an episodic phenomenon. Mov Disord. 2013 Sep 15;28(11):1509-19. doi: 10.1002/mds.25683. PMID 24132839
- [Background] Alice N, Fabienne C, Anne-Marie W, Kaat D. Does freezing in Parkinson's disease change limb coordination? A kinematic analysis. J Neurol. 2007 Sep;254(9):1268-77. doi: 10.1007/s00415-006-0514-3. Epub 2007 Apr 2. PMID 17401738
- [Background] Nieuwboer A, Dom R, De Weerdt W, Desloovere K, Fieuws S, Broens-Kaucsik E. Abnormalities of the spatiotemporal characteristics of gait at the onset of freezing in Parkinson's disease. Mov Disord. 2001 Nov;16(6):1066-75. doi: 10.1002/mds.1206. PMID 11748737
- [Background] Hausdorff JM, Schaafsma JD, Balash Y, Bartels AL, Gurevich T, Giladi N. Impaired regulation of stride variability in Parkinson's disease subjects with freezing of gait. Exp Brain Res. 2003 Mar;149(2):187-94. doi: 10.1007/s00221-002-1354-8. Epub 2003 Jan 22. PMID 12610686
- [Background] Siviy C, Baker LM, Quinlivan BT, Porciuncula F, Swaminathan K, Awad LN, Walsh CJ. Opportunities and challenges in the development of exoskeletons for locomotor assistance. Nat Biomed Eng. 2023 Apr;7(4):456-472. doi: 10.1038/s41551-022-00984-1. Epub 2022 Dec 22. PMID 36550303
- [Background] Macht M, Kaussner Y, Moller JC, Stiasny-Kolster K, Eggert KM, Kruger HP, Ellgring H. Predictors of freezing in Parkinson's disease: a survey of 6,620 patients. Mov Disord. 2007 May 15;22(7):953-6. doi: 10.1002/mds.21458. PMID 17377927
- [Background] Nutt JG, Bloem BR, Giladi N, Hallett M, Horak FB, Nieuwboer A. Freezing of gait: moving forward on a mysterious clinical phenomenon. Lancet Neurol. 2011 Aug;10(8):734-44. doi: 10.1016/S1474-4422(11)70143-0. PMID 21777828
- [Background] Jacobs JV, Nutt JG, Carlson-Kuhta P, Stephens M, Horak FB. Knee trembling during freezing of gait represents multiple anticipatory postural adjustments. Exp Neurol. 2009 Feb;215(2):334-41. doi: 10.1016/j.expneurol.2008.10.019. Epub 2008 Nov 12. PMID 19061889
- [Background] Mancini M, Shah VV, Stuart S, Curtze C, Horak FB, Safarpour D, Nutt JG. Measuring freezing of gait during daily-life: an open-source, wearable sensors approach. J Neuroeng Rehabil. 2021 Jan 4;18(1):1. doi: 10.1186/s12984-020-00774-3. PMID 33397401